CLINICAL TRIAL: NCT07321847
Title: Intratumoral Injection of IP-001 Following Standard-of-care Complete Hepatic Tumor Ablation in Patients With Liver-only Metastatic Colorectal Cancer
Brief Title: Injection of IP-001 Into Thermally Ablated Hepatic Tumors in Patients With Colorectal Liver Metastases
Acronym: INJECTABL-3
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Immunophotonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IP-IIO-925; 2025-524154-33-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-04; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer (CRC); Colon Cancer Liver Metastases; Rectal Cancer; Rectal Cancer With Liver Metastases; Colorectal Liver Metastasis (CRLM)
Keywords: Colorectal liver metastases; Colorectal cancer; Microwave ablation; Thermal ablation; Intratumoral immunotherapy; Intratumoral injection; Immune activation; Ablation-induced immunity; Liver tumor ablation; Metastatic cancer; Cancer; IP-001; Tumor ablation; Systemic immune response; Interventional immuno-oncology; Interventional oncology; Abscopal effect; T-cell stimulation
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — N-dihydrogalactochitosan; Injections; Water; Microwaves

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of three treatment arms. Each participant receives only the intervention assigned to their study arm, and there is no crossover between groups. The model is designed to evaluate whether adding IP-001 to the ablation procedure enhances local or systemic immune responses compared with ablation alone. All interventions are delivered in a single treatment session, and participants are followed prospectively for safety, feasibility, and early signals of antitumor activity.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: SOC CRLM ablation + 10 mg/mL IP-001 (IMP) (Experimental): SOC CRLM ablation: Standard of care microwave ablation is a procedure where a doctor uses imaging, such as ultrasound or CT, to guide a thin needle-like probe into a tumor. Once the probe is in place, it gives off microwave energy that heats the tumor from the inside. This heat destroys the cancer cells in that specific spot.
  10 mg/ml IP-001 (IMP): IP-001 is a study medication made from a type of sugar-based molecule designed to help the immune system recognize cancer cells. The 10 mg/mL means there are 10 milligrams of the medication in each milliliter of liquid. IP-001 is injected directly into the area that was treated with ablation, where it stays local and is meant to boost the body's immune response against the cancer.
  Interventions: Drug: 1.0% IP-001 for Injection, a 10 mg/mL solution of IP-001 in water; Procedure: Microwave (thermal) tumor ablation
- Arm 2: SOC CRLM ablation + 1 mg/mL IP 001 (Diluted IMP) (Experimental): SOC CRLM ablation: Standard of care microwave ablation is a procedure where a doctor uses imaging, such as ultrasound or CT, to guide a thin needle-like probe into a tumor. Once the probe is in place, it gives off microwave energy that heats the tumor from the inside. This heat destroys the cancer cells in that specific spot.
  1 mg/ml IP-001: IP-001 is a study medication made from a type of sugar-based molecule designed to help the immune system recognize cancer cells. The 1 mg/mL strength means the medication has been mixed with liquid so that there is 1 milligram of IP-001 in each milliliter of solution. This is a diluted version of the medication. IP-001 is injected directly into the area that was treated with ablation, where it stays local and is meant to boost the body's immune response against the cancer.
  Interventions: Drug: 1.0% IP-001 for Injection, a 1 mg/mL solution of IP-001 in water.; Procedure: Microwave (thermal) tumor ablation
- Control Arm: SOC CRLM ablation alone (Active Comparator): SOC CRLM ablation: Standard of care microwave ablation is a procedure where a doctor uses imaging, such as ultrasound or CT, to guide a thin needle-like probe into a tumor. Once the probe is in place, it gives off microwave energy that heats the tumor from the inside. This heat destroys the cancer cells in that specific spot.
  Interventions: Procedure: Microwave (thermal) tumor ablation

INTERVENTIONS:
Drug: 1.0% IP-001 for Injection, a 10 mg/mL solution of IP-001 in water — IP-001 is a novel, non-cytotoxic, immunostimulatory glycan polymer administered as a single intratumoral injection into the ablation zone immediately following standard of care image-guided microwave thermal ablation of a target tumor lesion.
  Other Names: IP-001
  Arms: Arm 1: SOC CRLM ablation + 10 mg/mL IP-001 (IMP)
Drug: 1.0% IP-001 for Injection, a 1 mg/mL solution of IP-001 in water. — IP-001 is a novel, non-cytotoxic, immunostimulatory glycan polymer administered as a single intratumoral injection into the ablation zone immediately following standard of care image-guided microwave thermal ablation of a target tumor lesion.
  Other Names: IP-001
  Arms: Arm 2: SOC CRLM ablation + 1 mg/mL IP 001 (Diluted IMP)
Procedure: Microwave (thermal) tumor ablation — Microwave ablation is a common medical procedure where doctors use imaging (like ultrasound or CT) to guide a thin probe into a tumor. The probe gives off microwave energy that heats up the tumor from the inside, causing the cancer cells in that spot to die.
  Unlike treatments such as chemotherapy or immunotherapy, which travel through the whole body, microwave ablation works only on the specific area being treated. It does not involve any drugs or medicines circulating in the bloodstream. It is a local treatment that targets just the tumor.
  Other Names: MWA; Microwave ablation; Microwave tumor ablation

SUMMARY:
The goal of this clinical trial is to learn if a new injectable drug (IP-001), administered after standard liver tumor ablation, can help prevent cancer from returning in people (males/females, ≥18 years old) with colorectal cancer that has spread only to the liver. The study will determine if injecting IP-001 into a liver tumor(s) after ablation will reduce the risk of cancer coming back in the liver and from spreading elsewhere in the body, will stimulate the immune system, will have any side effects, and will help improve a patient's response to other cancer therapies.

Researchers will compare a standard of care liver ablation alone (microwave ablation [MWA], a technique that destroys tumors using heat), with MWA plus a high-dose IP-001 or MWA with a low-dose IP-001. During the treatment procedures, the doctor first performs the standard microwave ablation to destroy the tumor. Then, in the experimental-drug arms, IP-001 is injected in and around the treated tumor area to activate the immune system locally so that the body is more likely to find and eliminate any remaining cancer cells.

DETAILED DESCRIPTION:
This is a Phase 2/3, three-arm, dose finding, randomized, controlled, patient-blinded, international, adaptive design study in patients with liver-only metastatic colorectal cancer. The purpose is to investigate the efficacy and safety of the two different dose concentrations of IP-001 for Injection administered intratumorally following standard of care (SOC) complete thermal ablation of liver tumors with microwave ablation (MWA) compared SOC MWA alone. MWA alone is selected as the control because, in patients with liver-only metastatic colorectal cancer treated with curative intent, MWA is an accepted SOC therapeutic strategy and routine continuation of systemic therapy in this context is not mandated by guidelines and remains heterogeneous across institutions.

The study is designed with a seamless transition from Phase 2 to the Phase 3 based on prespecified dose selection and interim efficacy and safety criteria. Phase 2 will include three-arms: MWA alone, MWA plus 10 mg/ml IP-001, or MWA plus 1 mg/ml IP-001. Crossover from the Control Arm to an Experimental Arm is not allowed. Phase 3 will continue to be randomized between the MWA alone (control) and the MWA plus IP-001 dose selected based on the Phase 2 interim (futility) analysis.

The trial will consist of the following three periods described below.

1. Screening Period: Up to 28 days for screening assessments to determine study eligibility.
2. Treatment and Follow-up Period: On Treatment Day 1, in a single session, all patients will undergo SOC hepatic tumor MWA with predetermined margins. Immediately following ablation, patients in the Experimental Arms will receive the appropriate dose of IP-001 intratumorally into all ablated tumor(s). Blood samples will be taken before treatment starts, and then again on various days after treatment to help check for important blood markers in and how the drug works in the body. In addition, patients will undergo post-treatment efficacy and safety and tolerability efficacy assessments for 12 weeks before patients move on to standard surveillance monitoring.
3. Surveillance Period: Patients will be followed for efficacy, concomitant medication and procedures, and survival, every 3 months for the first year, and then every 6 months thereafter for 5 years after the initial treatment.

Patients who develop a new or recurrent tumor(s) may be eligible receive additional treatment, as appropriate, including study retreatment, other standard liver treatments, or systemic anti-cancer therapy. Patients will be followed for subsequent anticancer therapies/procedures, progression, and survival status, as indicated, for 5 years after the original treatment day to help researchers determine if IP-001 will improve a patient's response to other cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 y of age at the time of signing the Informed Consent Form in accordance with local regulatory and/or national laws and International Council for Harmonisation (ICH)/Good Clinical Practice (GCP) regulations (consent must be received before any study-specific activity is performed).
2. Patients with liver-only metastatic CRC (and no radiologic or clinical evidence of extrahepatic metastases) with:

   1. No more than 5 CRLM (≤ 3 cm for largest diameter)
   2. An indication to receive percutaneous or laparoscopic SOC complete CRLM ablation with the intent of leaving no detectable liver disease
   3. Tumors amenable to ablation treatment in a single session
   4. No residual primary colorectal tumor at Treatment Day 1 or plans to have the primary tumor excised within 4-12 weeks following Treatment Day 1. (Patients with rectal cancer who underwent chemoradiotherapy for the primary cancer must have a complete clinical response.)
3. Prior systemic anticancer treatment for metastatic colorectal cancer is permitted but not required. Patients must have received no more than two prior lines of systemic anticancer treatment for mCRC.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 2.
5. Patients with adequate hematological function (defined as an absolute neutrophil count ≥ 1.5 × 109/L, hemoglobin level ≥ 9 g/dL, and platelet count ≥ 50 × 109/L) and coagulation function (defined as a partial thromboplastin time [PTT] or activated PTT [aPTT] and international normalized ratio [INR] ≤ 1.5 × the upper limit of normal [ULN]). (Note: the criteria for adequate hematological function must be met without erythropoietin dependency, use of growth factors, or the requirement for transfusions of blood, coagulation factors, platelets, or albumin within 14 d of Treatment Day 1.)
6. Patients with adequate hepatic function, defined as aspartate aminotransferase (AST) and alanine aminotransaminase (ALT) levels of ≤ 5 × the ULN, and a total bilirubin level ≤ 1.5 × the ULN (patients with documented Gilbert disease are allowed to participate in the study if their total bilirubin level is ≤ 3 × the ULN).
7. Patients with adequate renal function, defined as an estimated glomerular filtration rate (eGFR) ≥ 30 mL/min or an estimated creatinine clearance ≥ 40 mL/min (measured or calculated using the Cockcroft-Gault formula).
8. Women with childbearing potential (WOCBP)

   1. Must have a negative serum human chorionic gonadotropin pregnancy test in the Screening Period.
   2. Are using highly effective contraception, are not lactating, and agree not to become pregnant during the trial treatment period and for 187 days after treatment with the investigational drug.
9. Men agree not to donate sperm or to father a child during the trial treatment period and for 97 days after treatment with the investigational drug.

Exclusion Criteria:

1. Patients from vulnerable populations (incapacitated or unconscious individuals, persons deprived of liberty).
2. Patients with a known allergic reaction or hypersensitivity to shellfish, crabs, crustaceans, or any components used in trial treatment.
3. Patients with any prior treatment with IP-001 for Injection in a different clinical trial.
4. Patients who underwent any surgical liver resection, hepatic ablation or other hepatic locoregional therapy for CRLM within 3 months before Treatment Day 1; patients who received any other medical procedure, SACT, or treatment with any other investigational anticancer agents within 14 days before Treatment Day 1, or patients who at study enrollment have plans to receive SACT or locoregional therapies/procedures prior to intrahepatic or extrahepatic progression.
5. Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 d of randomization. Inhaled or topical steroids and adrenal replacement steroid doses (> 10 mg daily prednisone equivalent) are permitted in the absence of active autoimmune disease.
6. Patients who at screening have not recovered back to baseline or ≤ Grade 1 per National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) guidelines v6.0 from ongoing conditions related to any prior medicinal or procedural treatments (including major surgery) except for residual toxicities, unless conditions are deemed clinically non-significant by the Investigator and/or stable on supportive therapy (in consultation with Sponsor Medical Monitor), such as alopecia or Grade 2 neuropathy.
7. Patients with any extrahepatic nodal or non-nodal CRC metastases, except:

   1. History of infiltrated regional lymph nodes associated with the primary tumor if these lymph nodes were removed together with the primary tumor.
   2. Pulmonary nodules unless they are considered suspect for metastases because they show at least one of the following characteristics:

   i. new or increasing in size (at least 20% increase in longest diameter) in the last 12 mo; ii. unequivocal 18F-FDG tracer-uptake on PET; iii. solitary nodule >1 cm; iv. 2 - 5 nodules with at least 1 ≥ 0.8 cm; v. more than 5 nodules (excluding nodules that are stable in size over at least 1 y).
8. Patients with a history of another active malignancy within 2 years prior to Treatment Day 1, except for superficial skin cancers or localized, low-grade tumors deemed cured and not treated with systemic therapy. Patients with incidental prostate cancer may enroll if Stage ≤ T2N0M0 and Gleason score ≤ 6.
9. Patients with bleeding diathesis or anti-coagulation treatment that cannot be stopped 24 hours prior to Treatment Day 1 (low-dose aspirin will be allowed).
10. Patients who have one of the following cardiovascular disorders:

    1. Severe or uncontrolled cardiovascular disease (congestive heart failure New York Heart Association classification III or IV), or
    2. Unstable angina pectoris or a history of myocardial infarction within the last 6 mo, or
    3. Serious arrhythmias requiring medication (with the exception of atrial fibrillation or paroxysmal supraventricular tachycardia), or
    4. Significant QT-prolongation (QTcF ≥ 480 msec on screening electrocardiogram [ECG] [QTcF interval is not relevant in patients with pacemaker-controlled arrythmia]), or
    5. Uncontrolled hypertension, defined as a resting systolic blood pressure > 150 mmHg and/or resting diastolic blood pressure > 90 mmHg, which cannot be controlled by anti-hypertensive therapy.
11. Patients with any of the following infections/diseases:

    1. Known history of human immunodeficiency virus infection,
    2. Known active Hepatitis B or C viral infection,
    3. Any uncontrolled active systemic infection requiring intravenous antimicrobial treatment during screening,
    4. Any active, known, or suspected autoimmune disease.
12. Patients with a requirement for hemodialysis or peritoneal dialysis.
13. Patients with a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan or cavitating pulmonary lesion(s) or a known endobronchial disease manifestation.
14. Patients who received a live, attenuated vaccine within 28 days of Treatment Day 1.
15. Patients with any other serious underlying medical, psychological, familial, or geographical condition that, in the judgment of the Investigator, may limit compliance with the study or place the patient at high risk for treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 717 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2033-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy of IP-001 following standard-of-care (SOC) complete hepatic tumor ablation vs SOC complete hepatic tumor ablation alone in prolonging progression-free survival | From date of randomization to first documented progression (extrahepatic, or intrahepatic that could not be treated with curative-intent locoregional therapy) or death from any cause, whichever comes first, assessed up to 5 years.
  Progression-free survival (PFS) is defined as the time from randomization to first occurrence of objectively documented (1) extrahepatic progression or (2) intrahepatic progression (that could not be treated with curative-intent locoregional therapy) per RECIST v1.1, assessed by a Blinded Independent Central Review (BICR), or (3) death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
To compare disease control of IP-001 following SOC complete hepatic tumor ablation vs SOC complete hepatic tumor ablation alone | From date of randomization to first documented progression (extrahepatic, or intrahepatic that could not be treated with curative-intent locoregional therapy) or death from any cause, whichever comes first, assessed up to 5 years.
  * Extrahepatic PFS (ePFS) is defined as the time from randomization to first documented extrahepatic progression per RECIST v1.1 assessed by BICR, or death from any cause, whichever occurs first.
  * Intrahepatic PFS (iPFS) is defined as the time from randomization to first documented intrahepatic progression per RECIST v1.1 assessed by BICR, or death from any cause, whichever occurs first.
  * PFS is defined as the time from randomization to first documented (1) extrahepatic progression or (2) intrahepatic progression that could not be treated with curative-intent locoregional therapy per RECIST v1.1, assessed by the Investigator, or (3) death from any cause, whichever occurs first.
  * ePFS is defined as the time from randomization to first occurrence of objectively documented extrahepatic progression per RECIST v1.1, assessed by the Investigator, or death from any cause, whichever occurs first.
To compare survival outcomes of IP-001 following SOC complete hepatic tumor ablation vs SOC complete hepatic tumor ablation alone | From date of randomization to first documented progression (extrahepatic, or intrahepatic that could not be treated with curative-intent locoregional therapy) or death from any cause, whichever comes first, assessed up to 5 years.
  Overall survival (OS) is defined as the time from randomization to death from any cause.
To compare time to progression events between IP-001 following SOC complete hepatic tumor ablation and SOC complete hepatic tumor ablation alone | From date of randomization to first documented progression (extrahepatic or intrahepatic), assessed up to 5 years.
  * Time to Progression (TTP) is defined as the time from randomization to objectively documented intrahepatic or extrahepatic progression, per RECIST v1.1, assessed by BICR.
  * TTP is defined as the time from randomization to objectively documented intrahepatic or extrahepatic progression, per RECIST v1.1, assessed by the Investigator.
  * Time to Loss of Hepatic Control (TLHC) is defined as the time from randomization to objectively documented intrahepatic progression that cannot be treated with curative intent by locoregional therapy, assessed by the Investigator.
To compare safety and tolerability (via incidence of treatment-emergent adverse events) of IP-001 following SOC complete hepatic tumor ablation and SOC complete hepatic tumor ablation alone. | 12 weeks following treatment or resolution (whichever is longer).
  Incidence and severity of AEs, serious adverse events (SAEs), adverse events of special interest (AESIs), deaths, and laboratory abnormalities.
To compare the impact on patient-reported disease-specific health-related quality of life (HRQoL) outcomes of treatment with IP-001 following SOC complete hepatic tumor ablation vs SOC complete hepatic tumor ablation alone | From baseline (screening) until 1 year after treatment.
  Changes in questionnaire dimensions from baseline to 1 year post treatment as determined by scores on the patient-reported outcome (PRO) scale European Organization for the Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC) QLQ-C30 with the Colorectal Liver Metastases Module LMC21 for global health status/HRQoL, physical function, and role function.
To compare the impact on patient-reported general health-related quality of life (HRQoL) outcomes of treatment with IP-001 following SOC complete hepatic tumor ablation vs SOC complete hepatic tumor ablation alone | From baseline (screening) until patient's last visit, assessed up to 5 years.
  Changes in questionnaire dimensions from baseline to end of study as determined by scores on the patient-reported outcome (PRO) scale EuroQoL 5 Dimension 5 Level (EQ-5D-5L)
To determine the maximum plasma concentration (Cmax) of intratumorally administered IP-001 | Baseline (screening) through Day 45
  Cmax will be obtained after administration of IP-001
To determine the time to reach maximum plasma concentration (Tmax) of intratumorally administered IP-001 | Baseline (screening) through Day 45
  Tmax will be obtained after administration of IP-001
To determine the area under the plasma concentration-time curve (AUC0-t) of intratumorally administered IP-001 | Baseline (screening) through Day 45
  AUC0-t will be obtained after administration of IP-001
To determine the half-life (T1/2) of intratumorally administered IP-001 | Baseline (screening) through Day 45
  T1/2 will be obtained after administration of IP-001

CONTACTS AND LOCATIONS:
Overall Officials: Diane M Beatty, PhD, Study Director — Immunophotonics, Inc.

IPD SHARING:
Plan to Share IPD: No
No personal individual participant data will be shared (all data will be anonymized).